CLINICAL TRIAL: NCT00140660
Title: Randomized Study of ACVBP Versus ACVBP Plus Rituximab in Previously Untreated Patients Aged From 18 to 65 Years With Low-risk Localized Diffuse Large B-cell Lymphoma (Age-adjusted IPI = 0)
Brief Title: ACVBP Versus ACVBP Plus Rituximab in Low Risk Localized Diffuse Large B-cell Lymphoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low acrual
Sponsor: Lymphoma Study Association (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LNH03-1B
Record Dates: First submitted 2005-08-31; First posted 2005-09-01 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Diffuse Large Cell Lymphoma
Keywords: lymphoma, diffuse large B-cell; rituximab; chemotherapy
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- R-ACVBP (Experimental): addition of rituximab to standard ACVBP chemotherapy
  Interventions: Drug: rituximab
- ACVBP (No Intervention): standard ACVBP chemotherapy

INTERVENTIONS:
Drug: rituximab — 375 mg/m2 on D1
  Arms: R-ACVBP

SUMMARY:
This study is a multicentric randomized trial evaluating the efficacy of the combination R-ACVBP in patients 18 to 65 years with low risk localized diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
Approximately 30 to 40% of diffuse large B cell lymphomas are localized at diagnosis (stage I-II). Until the seventies, radiotherapy was used as the single modality to treat these localized stages but no more than half of the patients were cured. From the eighties, anthracycline-based regimens combined or not with radiotherapy gave superior results in term of relapse free survival compared with radiotherapy alone. Later on Miller et al. published a randomized study showing that 3 cycles of CHOP combined with radiotherapy gave superior results in term of overall survival as compared with 8 cycles of CHOP. This study was recently updated with a follow up of more than 8 years and shows no more difference between the two arms, due to an excess of late mortality after the combined treatment.

Recently, two trials were conducted by the GELA to compare chemotherapy alone to a combined chemo-radiotherapy approach in patients with low risk localized diffuse large cell lymphoma (age-adjusted IPI = 0).

* The objective of the LNH 93-1 study was to compare, in patients aged from 18 to 60 years 3 cycles of CHOP followed by radiotherapy with chemotherapy alone consisting in 3 cycles of ACVBP. The ACVBP regimen includes a more intensive induction followed by a sequential consolidation. With a median follow up of 55 months, the results have shown a superiority of the ACVBP arm for both the 5 year event free (83% vs. 74%, p = 0.004) and overall survival (89% vs. 80%, p = 0.02).
* The LNH 93-4 study compared in patients >60 years the association of 4 cycles of CHOP + radiotherapy to the same regimen without irradiation. This study fails to demonstrate any benefit of the combined chemo-radiotherapy in term of survival, but indicates that chemotherapy alone is probably less toxic in patients older than 69 years.

Considering these two trials, we concluded that radiotherapy given after chemotherapy did not give any benefit to elderly patients treated for a low risk localized diffuse large cell lymphoma, and that ACVBP regimen was superior to 3 CHOP + radiotherapy in patients <60 years, and has to be considered as the treatment of reference in these patients.

Two other GELA trials contributed recently to improve the treatment of diffuse large B cell lymphoma and have to be considered for the elaboration of future studies:

* The objective of the LNH 98-5 study was to compare the association of CHOP + rituximab (R-CHOP) to the CHOP regimen alone in elderly patients with previously untreated large B-cell lymphoma. The analysis showed a significant superiority of the association CHOP + rituximab.
* The LNH 93-5 study compared the ACVBP regimen to the CHOP in patients aged from 61 to 69 years with aggressive lymphoma and at least one adverse prognostic factor according to the International Prognostic Index. Out of 703 patients included in this study, the results have shown the same complete response rate in the two arms, but a significantly better 3-year event free survival and overall survival in the ACVBP arm than in the CHOP arm. However, the benefit seems to be greater in patients <66 years, due to higher toxicity with the ACVBP regimen in elderly patients.

All the above-mentioned results led us to propose a randomized trial comparing ACVBP to ACVBP + rituximab (R-ACVBP) in previously untreated patients with low risk localized diffuse large B-cell lymphoma (age-adjusted IPI = 0), and to extend the upper age limit from 60 to 65 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient with histologically proven CD20+ diffuse large B-cell lymphoma (WHO classification).
* Age from 18 to 65 years.
* Patient not previously treated.
* Ann Arbor stage I or II.
* ECOG performance status < 2.
* Normal LDH.
* Negative HIV, HBV and HCV serologies 4 weeks (except after vaccination).
* Having previously signed a written informed consent.

Exclusion Criteria:

* Any other histological type of lymphoma. vAny history of treated or non-treated indolent lymphoma. However, patients not previously diagnosed and having a diffuse large B-cell lymphoma with some small cell infiltration in lymph node may be included.
* Central nervous system or meningeal involvement by lymphoma.
* Contra-indication to any drug contained in the chemotherapy regimens.
* Poor renal function (creatinin level >150 mmol/l), poor hepatic function (total bilirubin level >30 mmol/l, transaminases >2.5 maximum normal level).
* Poor bone marrow reserve as defined by neutrophils < 1.5 G/l or platelets < 100 G/l.
* Any history of cancer during the last 5 years with the exception of non-melanoma skin tumors or stage 0 (in situ) cervical carcinoma.
* Any serious active disease (according to the investigator's decision).
* Treatment with any investigational drug within 30 days before planned first cycle of chemotherapy and during the study.
* Pregnant or lactating women
* Adult patient under tutelage.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2003-12 (Actual); Primary Completion 2008-07 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Event-free survival (EFS) | 4 years
  events defined as death from any cause, relapse for complete responders (CR) and unconfirmed complete responders (CRu), progression during and after treatment and change of therapy.

SECONDARY OUTCOMES:
Response rate at the end of the treatment | 6 months
Disease-free survival for complete responders | 4 years
Overall survival | 4 years
additionnal toxicities with R-ACVBP | 4 years
  number of SAE

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Ketterer, MD, Principal Investigator — Lymphoma Study Association; Felix Reyes, MD, Study Director — Lymphoma Study Association; Hervé Tilly, MD, Study Chair — Lymphoma Study Association; Corinne Haioun, MD, Study Chair — Lymphoma Study Association
Locations (11):
- Groupe d'Etude des Lymphomes de l'adulte, Mont-Godinne, Belgium
- France (9):
  - Hôpital Henri Mondor, Créteil
  - Hématologie CHU de Lille, Lille
  - Hôpital Saint Louis, Paris
  - Hématologie Adultes - Hôpital Necker, Paris
  - Service d'Hématologie - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Centre Hospitalier Robert Debré, Reims
  - Centre Henri Becquerel, Rouen
  - Hématologie CHU Purpan, Toulouse
  - Institut Gustave Roussy, Villejuif
- Centre Pluridisciplinaire d'Oncologie, CHUV, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reyes F, Lepage E, Ganem G, Molina TJ, Brice P, Coiffier B, Morel P, Ferme C, Bosly A, Lederlin P, Laurent G, Tilly H; Groupe d'Etude des Lymphomes de l'Adulte (GELA). ACVBP versus CHOP plus radiotherapy for localized aggressive lymphoma. N Engl J Med. 2005 Mar 24;352(12):1197-205. doi: 10.1056/NEJMoa042040. PMID 15788496
- [Background] Miller TP, Dahlberg S, Cassady JR, Adelstein DJ, Spier CM, Grogan TM, LeBlanc M, Carlin S, Chase E, Fisher RI. Chemotherapy alone compared with chemotherapy plus radiotherapy for localized intermediate- and high-grade non-Hodgkin's lymphoma. N Engl J Med. 1998 Jul 2;339(1):21-6. doi: 10.1056/NEJM199807023390104. PMID 9647875
- [Background] Feugier P, Van Hoof A, Sebban C, Solal-Celigny P, Bouabdallah R, Ferme C, Christian B, Lepage E, Tilly H, Morschhauser F, Gaulard P, Salles G, Bosly A, Gisselbrecht C, Reyes F, Coiffier B. Long-term results of the R-CHOP study in the treatment of elderly patients with diffuse large B-cell lymphoma: a study by the Groupe d'Etude des Lymphomes de l'Adulte. J Clin Oncol. 2005 Jun 20;23(18):4117-26. doi: 10.1200/JCO.2005.09.131. Epub 2005 May 2. PMID 15867204
- [Background] Tilly H, Lepage E, Coiffier B, Blanc M, Herbrecht R, Bosly A, Attal M, Fillet G, Guettier C, Molina TJ, Gisselbrecht C, Reyes F; Groupe d'Etude des Lymphomes de l'Adulte. Intensive conventional chemotherapy (ACVBP regimen) compared with standard CHOP for poor-prognosis aggressive non-Hodgkin lymphoma. Blood. 2003 Dec 15;102(13):4284-9. doi: 10.1182/blood-2003-02-0542. Epub 2003 Aug 14. PMID 12920037
- [Derived] Copie-Bergman C, Cuilliere-Dartigues P, Baia M, Briere J, Delarue R, Canioni D, Salles G, Parrens M, Belhadj K, Fabiani B, Recher C, Petrella T, Ketterer N, Peyrade F, Haioun C, Nagel I, Siebert R, Jardin F, Leroy K, Jais JP, Tilly H, Molina TJ, Gaulard P. MYC-IG rearrangements are negative predictors of survival in DLBCL patients treated with immunochemotherapy: a GELA/LYSA study. Blood. 2015 Nov 26;126(22):2466-74. doi: 10.1182/blood-2015-05-647602. Epub 2015 Sep 15. PMID 26373676
- See also: Official site of the Groupe d'Etudes des Lymphomes de l'Adulte (In french) — http://www.gela.org